CLINICAL TRIAL: NCT06759753
Title: Aleeto in Acute ISchemic Stroke：A RandomISed Controlled Clinical Trial
Acronym: ASSIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Executive Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HX-A-2024088
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
Keywords: Aleeto; Placebo parallel-controlled; Double Blind Study; Randomized Controlled Trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, double-blind, 1:1:1 randomized controlled study. 192 patients will be randomly assigned to 3 groups. Two dose groups are set 130μg/day and 260μg/day and one placebo group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental group 1 (Experimental): Intravenous administration of Aleeto at 130μg/day for 14±2 days (130μg Aleeto with 100 ml sodium chloride injection), along with Ginkgo Ester Dropping Pills, 4 pills per dose, 3 times/day, orally, for 90 days.
  Interventions: Drug: Aleeto
- Experimental group 2 (Experimental): Intravenous administration of Aleeto at 130μg/day for 14±2 days (260μg Aleeto with 100 ml sodium chloride injection), along with Ginkgo Ester Dropping Pills, 4 pills per dose, 3 times/day, orally, for 90 days.
  Interventions: Drug: Aleeto
- Placebo group (Placebo Comparator): Placebo with the same dosage form, odor and color as Aleeto was administered in the same way and course of treatment, along with Ginkgo Ester Dropping Pills, 4 pills per dose, 3 times/day, orally, for 90 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aleeto — According to the groups, patients would be treated with Aleeto via intravenous injection, and the specific dosage of Aleeto will depend on the grouping.
  Arms: Experimental group 1; Experimental group 2
Drug: Placebo — Placebo with the same dosage form, odor and color as Aleeto was administered in the same way and course of treatment.
  Arms: Placebo group

SUMMARY:
This study is a prospective, double-blind, 1:1:1 randomized controlled study aimed at evaluating the efficacy and safety of Aleeto treatment compared to placebo in improving the NIHSS score at 14 days in patients with moderate to severe acute ischemic stroke. It also aims to explore the neuroprotective effects of Aleeto in moderate to severe acute ischemic stroke and provide data support and evidence for future clinical trials and evidence-based medicine.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death worldwide, associated with high rates of morbidity, mortality, and disability. As a result, it places a significant social and economic burden on societies. Stroke is generally classified into two types: ischemic stroke and hemorrhagic stroke. Acute ischemic stroke (AIS) accounts for approximately 87% of all stroke cases, characterized by the sudden cessation of oxygen and blood supply to local cerebral tissue due to arterial occlusion.

According to the Global Burden of Disease study, in 2019, there were 28.76 million stroke patients in China, including 3.94 million new cases and 2.19 million deaths due to stroke. The burden of ischemic stroke (IS) in China has increased dramatically, with the Disability-Adjusted Life Years (DALYs) for IS rising by 138.6% from 1990 to 2019. This burden is expected to grow further due to the aging population, the persistently high incidence of stroke risk factors (such as hypertension), and inadequate management. Although significant advances have been made in the diagnosis and treatment of ischemic stroke in recent years-resulting in a notable reduction in recurrence rates-effective, targeted treatments to reduce disability and improve neurological recovery remain limited.

Aleeto, derived from cellular exosomes, is a group of specific protein polymers secreted by stem cells under stress. These exosomes possess several advantages, including selective assembly, targeted delivery, efficient tissue repair, high safety, stable chemical properties, and ease of preservation. Moreover, Aleeto has demonstrated strong potential for nerve repair.

This study is a single-center, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the safety, tolerability, and preliminary efficacy of Aleeto in patients with acute ischemic stroke. The trial also aims to determine the appropriate dosage for future clinical studies.

A total of 192 patients will be enrolled and randomly assigned to three groups. All participants will receive standardized treatment according to clinical guidelines, along with ginkgo ester dropping pills (4 pills per dose, 3 times per day, for 90 days of oral treatment). The dosage and type of drugs used will remain consistent throughout the trial.

Experimental Group 1: Intravenous administration of Aleeto at 130 μg/day for 14 ± 2 days (130 μg Aleeto dissolved in 100 mL sodium chloride injection).

Experimental Group 2: Intravenous administration of Aleeto at 260 μg/day for 14 ± 2 days (260 μg Aleeto dissolved in 100 mL sodium chloride injection).

Placebo Group: A placebo with the same appearance, odor, and color as Aleeto will be administered in the same manner and for the same duration as the experimental groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 30 and 80 years (30 ≤ age ≤ 80).
2. Diagnosis of acute ischemic stroke confirmed by CT or MRI, according to the "Key Points for Diagnosis of Major Cerebrovascular Diseases in China 2019."
3. Time from symptom onset ≤ 72 hours.
4. NIHSS score between 6 and 24, with a score of ≥ 1 on items 5 and 6 of the NIHSS.
5. Pre-stroke mRS (modified Rankin Scale) < 2, indicating independent activities of daily living.
6. Signed informed consent.

Exclusion Criteria:

1. Intracranial hemorrhagic diseases identified by head CT: cerebral hemorrhage, extradural hemorrhage, subarachnoid hemorrhage, intraventricular hemorrhage, etc.
2. Combined with other active and major neurological diseases (such as induced seizures, poor drug control of recurrent seizures, multiple sclerosis, intracranial tumors, etc.).
3. History of infectious diseases (HIV positive or positive test history, HCV antibody positive or positive test history, HBV surface antigen positive and/or serum HBV DNA positive or serum HBV DNA > 2 × 10^8 IU/ml).
4. Severe renal or hepatic insufficiency. (Severe hepatic insufficiency is defined as alanine aminotransferase (ALT) value>3 times normal upper limit or Aspartate aminotransferase (AST)>3 times normal upper limit; Severe renal insufficiency is defined as creatinine>1.5 times normal upper limit or creatinine clearance < 50 ml/min, or over stage 3 of chronic kidney disease), severe heart failure (New York Heart Association grades III - IV).
5. Resistant Hypertension, systolic pressure ≥220mmHg or diastolic pressure ≥120mmHg.
6. History of Hemostatic disorder, systemic bleeding, thrombocytopenia or neutropenia, drug-induced hematology or liver dysfunction, white blood cell count <2×10^9/L or platelet count <100×10^9/L.
7. History of severe anemia within the past 1 month (hemoglobin < 90g/L).
8. Body Mass Index (BMI) < 16kg/m2 or BMI> 35kg/m2.
9. Severe organic diseases with expected survival time <5 years, such as malignant tumor.
10. Women of child bearing potential, pregnant or breastfeeding.
11. Individual who have difficulty communicating verbally to the extent that they are unable to communicate, understand or follow instructions normally, and are unable to cooperate with treatment and evaluation.
12. Combined with alcohol and drug abuse history.
13. Known history of allergy to biological agents such as proteins and cell products.
14. History of intracranial or spinal surgery, major surgery, or severe physical trauma within the past 4 weeks.
15. Received any vaccinations within the past 28 days.
16. Use of other investigational drugs within 30 days or 5 drug half-lives.
17. Unable to complete follow-up due to geographical or other reasons.
18. The researchers believe that the patient is not suitable to participate in this study.
19. Participated in other clinical trials.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in NIH Stroke Scale | At 14 days after randomization
  NIH Stroke Scale (NIHSS) scores from 0 to 42. A higher score indicates worse neural function.

SECONDARY OUTCOMES:
Change from baseline in NIH Stroke Scale | At 7±1 days after randomization.
  NIH Stroke Scale (NIHSS) scores from 0 to 42. A higher score indicates worse neural function.
Change from baseline in Modified Rankin Scale | At 90±7days after randomization
  Modified Rankin Scale (mRS) ranks from 0 to 5. A higher rank indicates worse neural function.
Change from baseline in Fugl-Meyer Assessment | At 14±2 and 90±7days after randomization.
  Fugl-Meyer Assessment (FMA) socres from 0 to 226. A higher score indicates better motor function.
Change from baseline in Ashworth scale | At 14±2 and 90±7days after randomization.
  Ashworth scale ranks from 0 to 5. A higher rank indicates worse motor function.
The ratio of modified Barthel index ≥95 points | At 90±7days after randomization.
  Modified Barthel index socres from 0 to 100. A higher score indicates better self-care ability.
Change from baseline in Visual Analogue Scale | At 14±2 and 90±7days after randomization.
  Visual Analogue Scale (VAS) ranks from 0 to 10. A higher rank indicates higher pain level.
Change from baseline in Montreal Cognitive Assessment | At 90±7days after randomization.
  Montreal Cognitive Assessment (MoCA) socres from 0 to 30. A higher score indicates better cognitive function.
Combined vascular events | From randomization to the end of treatment at 90±7days
  Including stroke (including ischemic and hemorrhagic stroke), myocardial infarction and cardiovascular death
New-onset Stroke Events | From randomization to the end of treatment at 90±7days
  Including hemorrhagic and ischemic strokes
All-cause Mortality | From randomization to the end of treatment at 90±7 days

OTHER OUTCOMES:
Imaging markers of brain tissue edema | At 14±2 days post-randomization or before discharge
  Assessed by MRI Diffusion Tensor Imaging (DTI) and SPICE (SPectroscopic Imaging by exploiting Spatiospectral Correlation) rapid high-resolution 3D magnetic resonance spectroscopic imaging technique.
Neurocellular metabolic markers | At 14±2 days post-randomization or before discharge
  Assessed by MRI Diffusion Tensor Imaging (DTI) and SPICE (SPectroscopic Imaging by exploiting Spatiospectral Correlation) rapid high-resolution 3D magnetic resonance spectroscopic imaging technique.
Hypersensitivity events | From randomization to the end of treatment at 90±7days weeks
  Including skin reactions (rash, urticaria), eosinophilia, and one or more of the following: pulmonary lesions, hepatitis, tubular-interstitial nephritis, myocarditis, pericarditis, arthralgia, possibly accompanied by fever and lymphadenopathy
Serious adverse events | From randomization to the end of treatment at 90±7days weeks
  * Resulting in death
  * Immediately life-threatening(Life-threatening means that the event was immediately endangering the patient's life at the time it occurred, rather than the potential risk of death if the event worsens.)
  * Requires hospitalization or prolongation of hospitalization
  * Leads to lifelong or severe disability/functional impairment, or the loss of essential abilities to maintain normal daily living functions
  * Congenital anomalies, congenital defects, birth defects, or reproductive disorders
  * Major medical events that may endanger the subject, or require medical intervention to prevent any of the above outcomes.
Other adverse/serious adverse events | From randomization to the end of treatment at 90±7days weeks
  A. Laboratory tests: Safety tests include complete blood count, urine analysis, liver function, kidney function, coagulation, etc. Attention should be given to abnormal changes in laboratory results, and further testing may be required to assess their relevance to the study.
  B. Vital signs: The occurrence of abnormal temperature (≥38°C or ≤35°C), blood pressure (systolic BP ≥180 mmHg or <90 mmHg), respiratory rate (>24 breaths/min or other rhythm abnormalities), heart rate (>100 bpm or <60 bpm).

CONTACTS AND LOCATIONS:
Overall Officials: YiLong Wang, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No